CLINICAL TRIAL: NCT04112290
Title: A Prospective Incident Study of Arrhythmias in Hypertrophic Cardiomyopathy
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Jeffrey B. Geske, Principal Investigator, Mayo Clinic
Other Study IDs: 17-011376
Record Dates: First submitted 2019-09-28; First posted 2019-10-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Atrial fibrillation; Ventricular tachycardia; Arrhythmia; Hypertrophic cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Atrial Fibrillation; Tachycardia, Ventricular; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research study is to understand more about various heart rhythms (electrical problems) in persons with hypertrophic cardiomyopathy with and without sleep apnea.

DETAILED DESCRIPTION:
Adult patients with hypertrophic cardiomyopathy and without known atrial fibrillation or pacemaker/implantable cardiac defibrillation will undergo implantable loop recorder implantation. No direct interventions will be performed. Prospective observation of atrial and ventricular arrhythmia incidence and burden will be assessed, with additional analyses performed based on the presence or absence of obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Currently or previously enrolled in 17-003514 and 16-009474
* Adults age >18 years-old with a diagnosis of hypertrophic cardiomyopathy
* Both sexes
* Able to consent

Exclusion Criteria:

* Vulnerable study population
* Known atrial fibrillation or flutter (with the exception of post-operative atrial fibrillation)
* Pacemaker/ICD implantation
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with hypertrophic cardiomyopathy who are participating in (or previously participated in) Mayo Clinic study 17-003514 and/or 16-009474
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2019-11-05 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation incidence in hypertrophic cardiomyopathy | Final incidence to be calculated at study conclusion, after 3 years of rhythm monitoring.
  Define the incidence ratio of newly diagnosed atrial fibrillation in hypertrophic cardiomyopathy, with and without sleep apnea
Atrial fibrillation recurrence in hypertrophic cardiomyopathy | Final recurrence rate to be calculated at study conclusion, after 3 years of rhythm monitoring.
  Determine the frequency of recurrent atrial fibrillation in hypertrophic cardiomyopathy, with and without sleep apnea
Ventricular arrhythmia incidence in hypertrophic cardiomyopathy | Final incidence to be calculated at study conclusion, after 3 years of rhythm monitoring.
  Define the incidence ratio of newly diagnosed ventricular arrhythmias in hypertrophic cardiomyopathy, with and without sleep apnea

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Geske, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No